# SEQUENCED TREATMENT EFFECTIVENESS FOR POSTTRAUMATIC STRESS (STEPS)

## STATISTICAL ANALYSIS PLAN (SAP)

4/10/2024

## **Principal Investigator** John Fortney, PhD

## **Co-Principal Investigators**

Deborah Kaysen, PhD Charles Engel, MD, MPH

#### **Authors**

Brittany Blanchard, PhD Patrick Heagerty, PhD, John Fortney, PhD

## Supported by: Patient-Centered Outcomes Research Institute PTSD-2019C1-15636



**Modifications to the STEPS Statistical Analysis Plan** 

| Change | Reason | Date |
|---|---|---|
| Dropped "prefers<br>pharmacotherapy" from the list<br>of moderators examined. | Only 5.8% of respondents preferred pharmacotherapy over psychotherapy, which is too few to have sufficient power to test this hypothesis. | 6/21/24 |

## **Table of Contents**

| 1. | . Introduction | 4 |
|---|---|---|
| 2. | Study design | 4 |
| 3. | . Outcomes | 5 |
| 4. | Analyses | 6 |
| | 4.1. Primary, Secondary and Exploratory Outcomes (Hypotheses 1 and 2) | 6 |
| | 4.2 Moderation Analyses (Hypothesis 3) | 7 |
| 5. | Missing data | <u>9</u> |
| 6. | . Power and Sample Size Calculation | 9 |
| 7. | . References | 10 |
| 8. | Shell Tables and Figures | 11 |
| | Table S1. Baseline characteristics of patients enrolled in SPIRIT | 11 |
| | <b>Table S2.</b> Primary Outcomes: PTSD Symptom Severity Across Initial Treatment Arms | 17 |
| | Table S3. Secondary and Exploratory Outcomes Across Initial Treatment Arms | 18 |
| | Table S3. Secondary and Exploratory Outcomes Across Initial Treatment Arms, Continued | 19 |
| | Table S4. Primary Outcomes: PTSD Symptom Severity Across Sequenced Treatment Arms | 20 |
| | Table S6. Secondary and Exploratory Outcomes Across Sequenced Treatment Arms | 21 |
| | Table S6. Secondary and Exploratory Outcomes Across Sequenced Treatment Arms, continued | 24 |
| | Table S7. Main and Interaction effects of Moderators on Primary Outcome | 27 |

## 1. Introduction

Based on the state of the scientific evidence, the Sequenced Treatment Effectiveness for Posttraumatic Stress (STEPS) Trial was designed to address three specific aims. The first aim is to quantitatively compare engagement, self-reported PTSD symptom severity (primary outcome), quality of life, and recovery outcomes of primary care patients randomized to initially receive brief psychotherapy (Written Exposure Therapy - WET) or their choice of the three selective serotonin reuptake inhibitors (SSRIs). The second aim is, among patients not responding to initial treatment, to quantitatively compare outcomes of primary care patients randomized to: 1) augment the SSRI with WET, 2) switch from the SSRI to another class of antidepressants (serotonin-norepinephrine reuptake inhibitors - SNRI), or 3) switch from WET to the choice of the three SSRIs. The third specific aim is to quantitatively examine treatment heterogeneity among subgroups of primary care patients receiving pharmacotherapy and psychotherapy, including veterans, women, and those using cannabis.

This statistical analysis plan (SAP) will comprehensively enumerate the primary and secondary outcomes, moderating variables, and corresponding analyses.

## 2. Study design

As described in Figure 1, STEPS is a three-arm sequenced-treatment pragmatic trial.



Randomization – As depicted in Figure 1. Patients will initially be randomized to an SSRI (either sertraline, fluoxetine or paroxetine based on patient preference and treatment history) or Written Exposure Therapy (WET) in a 1:1 ratio. Randomization used randomly determined blocks sizes of 4, 6, or 8, and was stratified by healthcare system. Patients failing to respond to the initial treatment will receive the second treatment in the sequence.¹ Participants not responding to the SSRI in Arm 1 will have the SSRI augmented by WET. Participants not responding to the SSRI in Arm 2 will be switched from the SSRI to an SNRI (venlafaxine). Participants not responding to WET in Arm 3 will be switched from WET to an SSRI. The randomization scheme allocates patients not responding to treatment to these three sequenced treatments in a 1:1:2 ratio.

## 3. Outcomes

*Primary outcome*. The single primary outcome is PTSD symptom severity as measured by the PCL-5 (see Table 1).

Secondary outcomes. This study includes 6 secondary outcomes (Table 1). Secondary outcomes include health-related quality of life, recovery (not dominated by symptoms subscale), depression, anxiety, side-Effects, antidepressant discontinuation symptoms. Note that antidepressant discontinuation symptoms are only assessed for patients discontinuing an antidepressant and therefore we cannot compare this outcome across Arm 3 (WET) and Arms 1 and 2 (SSRI-SNRI and SSRI-WET). Therefore, this secondary outcome will only be reported descriptively for Arms 1 and 2.

*Exploratory outcomes*. This study includes 5 exploratory outcomes (Table 1). Secondary outcomes include treatment experiences, treatment engagement, clinical outcomes, recovery-oriented outcomes, and other outcomes.

Table 1. Outcome Survey Constructs, Instruments and Timeframes

| Construct/Instrument | Instruments | Eligibility<br>Assessment | Baseline | 4-<br>Month<br>Follow-<br>Up | 8-<br>Month<br>Follow-<br>Up |
|---|---|---|---|---|---|
| Primary Outcome | | | | | |
| PTSD Symptom Severity | PCL-5 | X | | Χ | Х |
| Secondary Outcomes | | | | | |
| Health-related Quality of Life | VR-12 | | Х | Χ | Х |
| Recovery, Not Dominated by<br>Symptoms | RAS, subscale | | Х | Х | Х |
| Depression | PHQ-9 | | Х | Х | Х |
| Anxiety | GAD-7 | | Х | Х | Х |
| Side-Effects | WFS | | Х | Х | Х |
| Antidepressant discontinuation symptoms | WFS | | Х | Х | Х |
| <b>Exploratory Outcomes</b> | | | | | |
| Alcohol Use | AUDIT-C | | Х | Χ | Х |

| Drug-Related Consequences | DAST-10 | Χ | Х | X |
|--------------------------------------|---------|---|---|---|
| Sleep | PSQI-A | Χ | Х | Χ |
| Service Utilization | WFS | Χ | Х | Х |
| Satisfaction with Mental Health Care | ECHO | Χ | Х | Х |
| Medication Adherence | WFS | Χ | Х | Х |

Note. AUDIT-C – Alcohol Use Disorder Identification Test – Concise; DAST-10 – Drug Abuse Screening Test; ECHO - Experience of Care & Health Outcomes; GAD-7 – Generalized Anxiety Disorder; PHQ-9 – Patient Health Questionnaire; PSQI-A - Pittsburgh Sleep Quality Index Addendum for PTSD; RAS – Recovery Assessment Scale VA – United States Department of Veterans Affairs; VR-12 – Veterans RAND 12-item Health Survey; WFS – Written for Study.

## 4. Analyses

## 4.1. Primary, Secondary and Exploratory Outcomes (Hypotheses 1 and 2)

- Aim 1: To quantitatively compare engagement, self-reported PTSD symptom severity (primary outcome), quality of life, and recovery outcomes of primary care patients randomized to initially receive brief psychotherapy (WET) or their choice of the three SSRIs.
  - Primary Hypothesis 1a Patients randomized to receive WET (Arm 3) will have better outcomes at 4 months than those randomized to an SSRI (Arms 1 and 2).

Data from the baseline and 4-month follow-up surveys will be used in the analysis. To account for potential intraclass correlation at the healthcare system level and the randomization stratified by healthcare system, healthcare system will be included as a fixed effect. Generalized linear models will be specified with the appropriate distribution and link functions, normal (linear), binary (logit), ordinal (logit), and count (Poisson/negative binomial depending on dispersion). The equation for a linear model is as follows:

$$Y_i = \beta_0 + \beta_1(WET\ Arm3) + C_i + e_i$$
(Eq. 1)

 $Y_i$  denotes the outcome (measured at 4 months) for individual i.  $\beta_0$  denotes the intercept. C denotes a vector of covariates (measured at baseline) that serve two functions: (1) dummy variables for healthcare systems to account for variation across systems as a fixed effect<sup>2</sup> and (2) additional baseline covariates and/or clinical outcomes theoretically related to both the outcome and the probability of missing follow-up surveys at 4-months. The effect of interest will be  $\beta_1$ , which represents the mean difference between SSRI (Arms 1 and 2) and WET (Arm 3) outcomes at 4 months. Table S2 presents a shell table for the primary outcome. Table S3 presents a shell table for the secondary and exploratory outcomes.

 Aim 2: For patients <u>not responding to initial treatment by 4 months</u>, to quantitatively compare engagement, self-reported PTSD symptom severity (primary outcome), quality of life, and recovery outcomes at 8 months of primary care patients randomized to: 1) switch from brief psychotherapy (WET) to their choice of the three SSRIs, 2) augment the SSRI with brief psychotherapy (WET), or 3) switch from one class of antidepressants (SSRI) to another class of antidepressants (SNRI - venlafaxine).

- Primary Hypotheses 2a Patients not responding to initial SSRI treatment, randomized to an SSRI <u>augmented</u> by WET (Arm 1) will have better outcomes at 8-months than those randomized to <u>switching</u> from an SSRI to an SNRI (Arm 2).
- Exploratory Hypotheses 2b Patient not responding to initial treatment randomized to an SSRI <u>augmented</u> by WET (Arm 1) will have better outcomes at 8-months than those randomized to <u>switching</u> from WET to their choice of the three SSRIs (Arm 3).

Data from the baseline and 8-month follow-up surveys will be used in the analysis, with the subset of patients not responding to the initial treatment. Otherwise, the analytical models will be specified the same as for Aim 1. There will be two models estimated represented by equation 2. The first model represents the comparison between Arm 1 (SSRI Augmented with WET) and Arm 2 (switched to SNRI). The second model represents the comparison between Arm 1 (SSRI augmented with WET) and Arm 3 (WET switched to SSRI). Table S4 presents a shell table for the primary outcome. Table S5 presents a shell table for the secondary and exploratory outcomes. The equation for a linear model is as follows:

$$Y_i = \beta_0 + \beta_1 (SSRI \ Augment \ WET \ Arm \ 1) + C_i + e_i$$
 (Eq. 2)

Effect sizes. Effect sizes will be reported for all outcomes. Cohen's *d* effect sizes will be calculated and presented with 95% confidence intervals. Between group effect sizes will be calculated as the model-estimated treatment effect divided by the pooled, raw baseline standard deviation.

Statistical tests. Statistical tests will be only be conducted for the primary outcome (PCL-5). There will be a single hypothesis test for hypothesis 1a involving 4-month outcomes for the entire sample, and a single separate hypothesis for hypothesis 2a involving 8-month outcomes among those not responding to the initiation SSRI treatment.

## 4.2 Risk Factor and Treatment Moderator Analyses (Hypothesis 3)

Risk Factors. The following risk factors for poor outcomes will be examined (see Table 2): veteran status, combat exposure (reported as the most bothersome trauma), benzodiazepines use, current antidepressant use at baseline, and drug problems.

Treatment Moderators. The following moderators will be examined in the treatment heterogeneity analysis (see Table 2): Male gender, poor access, and cannabis use.

Table 2. Risk Factors and Treatment Moderator Survey Constructs, Instruments and Timeframes

| Construct/Instrument | Instruments | Eligibility<br>Assessment | Baseline | 4-<br>Month<br>Follow-<br>Up | 8-<br>Month<br>Follow-<br>Up |
|---|---|---|---|---|---|
| Risk Factors | | | | | |
| Veteran status (for FQHC patients) | WFS | | Χ | | |
| Combat Trauma Exposure | STQ <sup>3</sup> | Х | | | |
| Benzodiazepines Use | BAM-R <sup>4,5</sup> | | Х | | |
| Current Antidepressant Use | WFS | | Х | | |
| Drug Problems | DAST-10 <sup>6</sup> | | Х | | |
| Treatment Moderators | | | | | |
| Gender | WFS | | Х | | |
| Perceived Access to Mental Health | APAC <sup>7</sup> | | Х | | |
| Care | | | | | |
| Cannabis Use | WFS† | | Х | | |

<sup>†</sup> Only asked in states were cannabis use is legal

*Note.* APAC – BAM-R - Brief Addiction Monitor Revised; DAST-10 – Drug Abuse Screening Test; STQ – Short Trauma Questionnaire (first part of Posttraumatic Diagnostic Scale for DSM-5).

- Aim 3: To quantitatively examine treatment heterogeneity among subgroups of primary care patients receiving pharmacotherapy and psychotherapy.
  - Primary Hypothesis 3a: Improvements in PTSD symptom severity at 4-months will be less for: 1) veterans compared with non-veterans (adjusting for gender), 2) those with combat exposure (adjusting for gender) compared with other types of traumas, 3) those currently prescribed benzodiazepines, 4) those taking SSRIs/SNRIs at study entry, and 5) those with self-reported alcohol use and drug-related consequences.
  - Primary Hypothesis 3b: Male gender, poor access, and cannabis use will be treatment moderators of 4-month outcomes that reduce the differential effectiveness of psychotherapy compared to pharmacotherapy.

Risk factor main effects (Hypothesis 3a) will be evaluated jointly using the same model as described for the primary outcome (Equation 1). The equation for a linear model is as follows:

$$Y_i = \beta_0 + \beta_1 (Arm3 - WET) + \beta_2 R_i + C_i + e_i$$
 (Eq. 3)

 $R_i$  denotes a vector of risk factors (measured at baseline) for individual *i*. The effect of interest for hypothesis 3a will be  $\beta_2$ . Table S7 presents a shell table for the primary outcome.

Treatment moderator main effects (Hypothesis 3a) and interaction effects (Hypothesis 3b) will be tested jointly using the same model as described for the primary outcome (Equation 1). All moderators will be grand mean centered. The equation for the analytical model is as follows:

$$Y_i = \beta_0 + \beta_1 (Arm3 - WET) + \beta_2 M_i + \beta_3 (M_i \times (Arm3 - WET)) + C_i + e_i$$
(Eq. 4)

 $M_i$  denotes a vector of moderators (measured at baseline) for individual *i*.  $\beta_1$ , represents the main effect of the moderator. The effect of interest for hypothesis 3b will be  $\beta_3$ , which represents the interaction effect of the moderators as a group with the initial treatment group assignment. Table S7 presents a shell table for the primary outcome.

## 5. Missing data

Estimates from the models are unbiased under conditions of *Missing at Random* (MAR), which means that the mechanism of missingness is observed in the data. Most relevant to the current analysis, estimates will be unbiased when missingness is caused by previously observed values of the dependent variable, but not if missingness is caused by the unobserved value at the missing wave. For missing data, we will use multiple imputation with auxiliary variables. We will also attempt to make the MAR assumption more plausible by incorporating correlates with the reasons for missingness into the model.<sup>8</sup>

## 6. Power and Sample Size Calculation

With 350 patients randomized to pharmacotherapy (Arms 1 & 2) and 350 randomized to psychotherapy (Arm 3) and assuming a 20% attrition rate and α significance level of 0.05, we will have 80% power for Hypothesis 1 to detect mean differences of 0.24 standard deviations (effect size), or 4.08 points on the PCL-5 our primary outcome. With 175 patients in each arm, and conservatively assuming a 40% treatment non-response rate, and 20% attrition rate, we will have 80% power for Hypothesis 2a to detect means differences of 0.47 standard deviations, or 7.99 points for the PCL-5 score. For the heterogeneity analyses of current versus no SSRI/SNRI use at baseline we will have 80% power to detect differences in treatment effects comparing those subjects with and without SSRIs at baseline of 0.52, 0.48 and 0.47 standard deviations depending on the proportion of patients not taking SSRIs at study entry (30%, 40% or 50%). Assuming that 30% of patients are not taking SSRIs/SNRIs at study entry, we will have 80% power to detect difference in treatment effects of 8.84 on the PCL-5. Because we would have more power to detect treatment heterogeneity if 50% of patients were taking SSRIs/SNRIs at baseline, we now propose to prioritize enrollment of patients not taking SSRIs/SNRIs. If 50% of patients were taking SSRIs/SNRIs at baseline, we will have 80% power to detect differences in treatment effects of 7.99 on the PCL-5.

## 7. References

- 1. Stein D, Ipser J, Seedat S, Sager C, Amos T. Pharmacotherapy for post traumatic stress disorder (PTSD). *Cochrane Database of Systematic Reviews*. 2006(1).
- 2. McNeish D, Stapleton LM. Modeling Clustered Data with Very Few Clusters. *Multivariate behavioral research*. 2016;51(4):495-518.
- 3. Foa EB, McLean CP, Zang Y, et al. Psychometric properties of the Posttraumatic Diagnostic Scale for DSM-5 (PDS-5). *Psychological assessment.* 2016;28(10):1166-1171.
- 4. Hallinan S, Gaddy M, Ghosh A, Burgen E. Factor structure and measurement invariance of the Revised Brief Addiction Monitor. *Psychological assessment*. 2021;33(3):273-278.
- 5. Liebmann EP, Resnick SG, Hoff RA, Katz IR. Associations between patient experience and clinical outcomes in substance use disorder clinics: Findings from the veterans outcomes assessment survey. *Journal of substance abuse treatment*. 2022;133:108505.
- 6. Yudko E, Lozhkina O, Fouts A. A comprehensive review of the psychometric properties of the Drug Abuse Screening Test. *Journal of substance abuse treatment*. 2007;32(2):189-198.
- 7. Fortney JC, Pyne JM, Hawrilenko M, et al. Psychometric Properties of the Assessment of Perceived Access to Care (APAC) Instrument. *The Journal of ambulatory care management*. 2020.
- 8. Little RJ, D'Agostino R, Cohen ML, et al. The prevention and treatment of missing data in clinical trials. *The New England journal of medicine*. 2012;367(14):1355-1360.

## 8. Shell Tables and Figures

## **Table S1.** Baseline characteristics of patients enrolled in SPIRIT

| | Overall (N = 700) | Arm 1 (n = 179) | Arm2 (n = 169) | Arm3 (n = 352) |
|---|---|---|---|---|
| | N(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) |
| Socio-Demographic Characteristics | | | | |

#### Age

Ethnicity

Hispanic or Latina/o/e Not Hispanic or Latina/o/e Missing

Race and Ethnicity

American Indian, Alaskan Native, or other Indigenous group

Arab or Middle Eastern

Asian

Black or African American

Multi-race

Native Hawaiian or Pacific Islander

White

Another identity

Missing

#### Gender

Man

Woman

Transgender Man

Transgender Woman

Non-binary or gender fluid

Another identity

Missing

| Overall (N = 700) | Arm 1 (n = 179) | Arm2 (n = 169) | Arm3 (n = 352) |
|-------------------|-----------------|----------------|----------------|
| N(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) |

Sexual Orientation

Bisexual

Lesbian or gay

Straight or heterosexual

Another identity

Missing

#### Marital Status

Divorced

Married/Living with partner

Separated

Single, never married

Widowed

Missing

#### Education

<= 8<sup>th</sup> grade

Some high school

High school graduate

Some college

College graduate

Any postgraduate work

Missing

#### Veteran Status

No

Yes

Missing

## Employment

Full-time

Part-time

Temporarily laid off/on-strike

Unemployed

| Overall (N = 700) | Arm 1 (n = 179) | Arm2 (n = 169) | Arm3 (n = 352) |
|-------------------|-----------------|----------------|----------------|
| N(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) |

Retired

Disabled

Student

Missing

## **Household Poverty**

Above

Below

Missing

## Health Insurance<sup>1</sup>

Uninsured

Medicaid

Medicare

**Government Insurance** 

Private Insurance

Missing

## Endorsed and Anticipated Stigma Inventory (EASI)

Beliefs About Mental Health Treatment (range: 8-40)

Perceived Access to Mental Health Care (APAC) (range: 1-5)

Social Support (ESSI)

Low Social Support (ESSI <= 18)

High Social Support (ESSI > 18)

Missing

Number of people that can give you support

Health Literacy Screener (range: 3-15)

Home Internet Access on Computer

Yes

No

Missing

| Overall (N = 700) | Arm 1 (n = 179) | Arm2 (n = 169) | Arm3 (n = 352) |
|-------------------|-----------------|----------------|----------------|
| N(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) |

#### **Clinical Characteristics**

```
Perceived need for treatment (NCS-R)
Yes
No
Missing

Treatment history (NCS-R)
Past use of psychotropic medication
Yes
No
```

Age first used psychotropic medication

Past use of psychotherapy

Yes

No

Missing

Missing

Age at first psychotherapy session

## Currently taking antidepressant<sup>1</sup>

No

Yes, Sertraline

Yes, fluoxetine

Yes, paroxetine

Yes, venlafaxine

Yes, citalopram

Yes, escitalopram

Yes, duloxetine

Yes, bupropion

Missing

Most Bothersome Trauma (Short Trauma Questionnaire)

Serious Life Threatening Illness

**Physical Assault** 

| Overall (N = 700) | Arm 1 (n = 179) | Arm2 (n = 169) | Arm3 (n = 352) |
|-------------------|-----------------|----------------|----------------|
| N(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) |

Sexual Assault

Military combat or lived in a war zone

Child Abuse

Accident

Natural Disaster

Other

Missing

Treatment Acceptability

Medication Acceptability

**Definitely Not Acceptable** 

Probably Not Acceptable

Probably Acceptable

**Definitely Acceptable** 

Missing

Psychotherapy Acceptability

**Definitely Not Acceptable** 

Probably Not Acceptable

Probably Acceptable

**Definitely Acceptable** 

Missing

Short Form (VR12)

Physical Health Component Summary (range: 0-100)

#### Outcomes

PTSD Checklist (PCL-5) (range: 0-80)

Short Form (VR12)

Mental Health Component Summary (range: 0-100)

Recovery Assessment Scale (RAS)

Not dominated by symptoms (range: 1-5)

| | Overall (N = 700) | Arm 1 (n = 179) | Arm2 (n = 169) | Arm3 (n = 352) |
|---|---|---|---|---|
| | N(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) | n(%) or μ(SD) |
| Patient Health Questionnaire (PHQ-9) (range: 0-27) | | | | |

Generalized Anxiety (GAD-7) (range: 0-21)

Sleep (PSQI-A) (range: 0-21)

Alcohol Use (AUDIT) (range: 0-12)

Number of days using cannabis in the past 30 days

Not Applicable<sup>2</sup>
On days using cannabis, how many times using per day

Not Applicable<sup>2</sup>

Drug Use (DAST-10)

No drug use

Low level (1-2)

Moderate level (3-5)

Substantial level (6-8)

Severe level (6-8)

Missing

#### Side Effects

Average number of 'Often' or 'Always' responses to being bothered by side effects in the past 30 days

Not Applicable (not currently taking psychotropic medication)

1. Not mutually exclusive

**Table S2.** Primary Outcomes: PTSD Symptom Severity Across Initial Treatment Arms

| | | Arms 1 an | d 2 (SSRI) | Arm 3 | (WET) | Difference in Treatment Arr | | nt Arms |
|---|---|---|---|---|---|---|---|---|
| PCL-5 | No. | Mean (SD) | 95% CI | Mean (SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Baseline | | | | | | - | ı | - |
| 4-Months | | | | | | | | |

**Table S3.** Secondary and Exploratory Outcomes Across Initial Treatment Arms

| | | Arms 1 ar | nd 2 (SSRI) | Arm 3 (WET) | | Difference in Treatment Arms | | |
|---|---|---|---|---|---|---|---|---|
| Secondary Outcomes | No. | Mean<br>(SD) | 95% CÍ | Mean<br>(SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Mental Health-related<br>Quality of Life | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | | | |
| Recovery, Not Dominated by Symptoms | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | | | |
| Depression | | | | | | | | |
| Baseline | | | | | | - | _ | - |
| 4-Months | | | | | | | | |
| Anxiety | | | | | | | | |
| Baseline | | | | | | _ | - | - |
| 4-Months | | | | | | | | |
| Side-Effects | | | | | | | | |
| Baseline | | | | | | - | _ | - |
| 4-Months | | | | | | | | |
| Antidepressant discontinuation symptoms | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | | | |

**Table S3.** Secondary and Exploratory Outcomes Across Initial Treatment Arms, Continued

| | | Arms 1 aı | Arms 1 and 2 (SSRI) | | Arm 3 (WET) | | Difference in Treatment Arms | |
|---|---|---|---|---|---|---|---|---|
| Exploratory Outcomes | No. | Mean<br>(SD) | 95% Ci | Mean<br>(SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Alcohol Use | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | | | |
| Drug Problems | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | | | |
| Sleep | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | | | |
| Service Utilization | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | | | |
| Satisfaction with Mental<br>Health Care | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | | | |
| Treatment Engagement | | | | | | | | |
| 4-Months | | | | | | | | |

**Table S4.** Primary Outcomes: PTSD Symptom Severity Across Sequenced Treatment Arms

| | | Arr | n 1 | Arr | n 2 | Differer | Difference in Treatment Arms | |
|---|---|---|---|---|---|---|---|---|
| | | (Augment | SSRI-WET) | (Switch S | SRI-SNRI) | | | |
| PCL-5 | No. | Mean (SD) | 95% CI | Mean (SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| | | Arn<br>(Augment | | Arr<br>(Switch V | n 3<br>VET-SSRI) | Difference in Treatment Arms | | |
| | No. | Mean (SD) | 95% CI | Mean (SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |

**Table S6.** Secondary and Exploratory Outcomes Across Sequenced Treatment Arms

| | | | Arm 1<br>(Augment SSRI-WET) | | Arm 2<br>(Switch SSRI-SNRI) | | Difference in Treatment Arms | |
|---|---|---|---|---|---|---|---|---|
| Secondary Outcomes | No. | Mean (SD) | 95% CI | Mean (SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Mental Health-related | | | | | | | | |
| Quality of Life | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | = | - |
| 8-Months | | | | | | | | |
| Recovery, Not Dominated | | | | | | | | |
| by Symptoms | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| Depression | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| Anxiety | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |

| Baseline | | | | | | - | - | - |
|---|---|---|---|---|---|---|---|---|
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| Antidepressant | | | | | | | | |
| discontinuation symptoms | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| | | | m 1 | | m 3 | Difference in Treatment Arms | | |
| | | | SSRI-WET) | (Switch V | VET-SSRI) | | | |
| | No. | Mean (SD) | 95% CI | Mean (SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Mental Health-related | | | - | | | Ρ | | <u> </u> |
| Quality of Life | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| Recovery, Not Dominated | | | | | | | | |
| by Symptoms | <del> </del> | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | <u> </u> | | | | | - | - | - |
| 8-Months | <del> </del> | | | | | | <del> </del> | _ |
| Depression | <u> </u> | | | | | | | |
| Baseline | <u> </u> | | | | | _ | _ | _ |
| Daseille | | | | | | - | | |

Side Effects

| 4-Months | - | - | - |
|--------------------------|---|---|---|
| 8-Months | | | |
| Anxiety | | | |
| Baseline | - | - | - |
| 4-Months | - | - | - |
| 8-Months | | | |
| Side Effects | | | |
| Baseline | - | - | - |
| 4-Months | - | - | - |
| 8-Months | | | |
| Antidepressant | | | |
| discontinuation symptoms | | | |
| Baseline | - | - | - |
| 4-Months | - | - | - |
| 8-Months | | | |

**Table S6.** Secondary and Exploratory Outcomes Across Sequenced Treatment Arms, continued

| | | Arm 1 | | Arr | n 2 | Difference in Treatment Arms | | |
|---|---|---|---|---|---|---|---|---|
| | | (Augment | SSRI-WET) | (Switch S | SRI-SNRI) | | | |
| Exploratory Outcomes | No. | Mean (SD) | 95% CI | Mean (SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Alcohol Use | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| Drug Problems | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| Sleep | | | | | | | | |
| Baseline | | | | | | - | - | _ |
| 4-Months | | | | | | - | - | - |
| 8-Months | | | | | | | | |
| Service Utilization | | | | | | | | |
| Baseline | | | | | | - | - | - |
| 4-Months | | | | | | - | - | _ |
| 8-Months | | | | | | | | |
| Satisfaction with Mental | | | | | | | | |
| Health Care | | | | | | | | |

| Desalina | | 一 | 1 | T 7 | | | | |
|---|---|---|---|---|---|---|---|---|
| Baseline | | | <del> </del> | <u> </u> | <del> </del> | - | - | - |
| 4-Months | | | <del> </del> | <u> </u> ' | <u> </u> | - | - | - |
| 8-Months | | | <del> </del> | | | | | <u> </u> |
| | | | 1 | ' | | | · | |
| Treatment Engagement | | | 1 | ' | | | | |
| 4-Months | | | <u> </u> | | | - | - | - |
| 8-Months | | | | ' | | | | ſ <u></u> ' |
| | | | 1 | | | | · | |
| | | Arn | n 1 | Arr | m 3 | Differen | nce in Treatme | nt Arms |
| | | (Augment S | SSRI-WET) | (Switch V | WET-SSRI) | | | |
| | No. | Mean (SD) | 95% CI | Mean (SD) | 95% CI | Adjusted<br>Group<br>Difference,<br>β | 95% CI | Cohen's d |
| Alcohol Use | | | 1 | 1 | | | | |
| Baseline | | | 1 | 1 | | - | - | - |
| 4-Months | | | 1 | <u> </u> | | - | - | - |
| 8-Months | | | 1 | ' | | | · | |
| Drug Problems | | | 1 | | | | | |
| Baseline | | | 1 | ' | | - | - | - |
| 4-Months | | | 1 | <u> </u> | | - | - | |
| 8-Months | | | 1 | ' | | | | |
| | | | 1 | | | | | |
| Sleep | | | 1 | 1 | | | | |
| Baseline | | | 1 | <u> </u> | | - | - | - |
| 4-Months | | <u> </u> | 1 | ' | | - | - | - |
| 8-Months | | | 1 | 1 | | | | |
| | | | 1 | 1 | | | | |
| Service Utilization | | <u> </u> | | | | | | |
| 4-Months 8-Months Drug Problems Baseline 4-Months 8-Months Sleep Baseline 4-Months 8-Months | | | | | | | - | - |

| Baseline | - | - | - |
|--------------------------|---|---|---|
| 4-Months | - | - | _ |
| 8-Months | | | |
| Satisfaction with Mental | | | |
| Health Care | | | |
| Baseline | - | - | - |
| 4-Months | - | - | - |
| 8-Months | | | |
| Treatment Engagement | | | |
| 4-Months | _ | - | - |
| 8-Months | | | |

**Table S7.** Main Effects of Risk Factors and Interaction Effects of Moderators on Primary Outcome

| | Main Effect | | Treatment Arm 3 (WET) Interaction | |
|---|---|---|---|---|
| | В | р | В | р |
| Risk Factors | | | | |
| Veteran status | | | - | - |
| Combat Trauma Exposure | | | = | - |
| Benzodiazepines Use | | | - | - |
| Current Antidepressant Use | | | - | - |
| Drug Problems | | | - | - |
| Treatment Moderator | | | | |
| Gender | | | | |
| Perceived Access to Mental | | | | |
| Health Care | | | | |
| Cannabis Use | | | | |
| Medication Acceptability > | | | | |
| Therapy Acceptability | | | | |